CLINICAL TRIAL: NCT01622673
Title: A Study to Evaluate the Effect of Metal Cation-Containing Antacids on Raltegravir Pharmacokinetics in HIV-Infected Subjects on a Stable Raltegravir-Containing Regimen
Brief Title: A Pharmacokinetic Study to Evaluate the Effect of Antacids on Raltegravir (MK-0518) in HIV-Infected Participants (MK-0518-247)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0518-247
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Results first posted 2013-09-17 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; aluminum hydroxide, magnesium hydroxide, simethicone drug combination; Magnesium; Aluminum Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- RAL, TUMS+RAL, MINTOX+RAL, MINTOX Before RAL, MINTOX After RAL (Experimental): Participants received Raltegravir in treatment period 1, followed by TUMS® + Raltegravir in treatment period 2, followed by MINTOX® + Raltegravir in treatment period 3, followed by MINTOX® 2 hours before Raltegravir in treatment period 4, followed by MINTOX® 2 hours After Raltegravir in treatment period 5. There was a 2-day washout between treatment periods.
  Interventions: Drug: Raltegravir; Drug: TUMS® Ultra Strength; Drug: MINTOX® Maximum Strength
- TUMS+RAL, MINTOX+RAL, RAL, MINTOX Before RAL, MINTOX After RAL (Experimental): Participants received TUMS® + Raltegravir in treatment period 1, followed by MINTOX® + Raltegravir in treatment period 2, followed by Raltegravir in treatment period 3, followed by MINTOX® 2 hours before Raltegravir in treatment period 4, followed by MINTOX® 2 hours after Raltegravir in treatment period 5. There was a minimum 2-day washout between treatment periods.
  Interventions: Drug: Raltegravir; Drug: TUMS® Ultra Strength; Drug: MINTOX® Maximum Strength
- MINTOX+RAL, RAL, TUMS+RAL, MINTOX Before RAL, MINTOX After RAL (Experimental): Participants received MINTOX® + Raltegravir in treatment period 1, followed by Raltegravir in treatment period 2, followed by TUMS® + Raltegravir in treatment period 3, followed by MINTOX® 2 hours before Raltegravir in treatment period 4, followed by MINTOX® 2 hours after Raltegravir in treatment period 5. There was a minimum 2-day washout between treatment periods.
  Interventions: Drug: Raltegravir; Drug: TUMS® Ultra Strength; Drug: MINTOX® Maximum Strength
- RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL (Experimental): Participants received Raltegravir in treatment period 1, followed by MINTOX® + Raltegravir in treatment period 2, followed by TUMS® + Raltegravir in treatment period 3, followed by MINTOX® 2 hours after Raltegravir in treatment period 4, followed by MINTOX® 2 hours before Raltegravir in treatment period 5. There was a minimum 2-day washout between treatment periods.
  Interventions: Drug: Raltegravir; Drug: TUMS® Ultra Strength; Drug: MINTOX® Maximum Strength
- TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL (Experimental): Participants received TUMS® + Raltegravir in treatment period 1, followed by Raltegravir in treatment period 2, followed by MINTOX® + Raltegravir in treatment period 3, followed by MINTOX® 2 hours after Raltegravir in treatment period 4, followed by MINTOX® 2 hours before Raltegravir in treatment period 5. There was a minimum 2-day washout between treatment periods.
  Interventions: Drug: Raltegravir; Drug: TUMS® Ultra Strength; Drug: MINTOX® Maximum Strength
- MINTOX+RAL, TUMS+RAL, RAL, MINTOX After RAL, MINTOX Before RAL (Experimental): Participants received MINTOX® + Raltegravir in treatment period 1, followed by TUMS® + Raltegravir in treatment period 2, followed by Raltegravir in treatment period 3, followed by MINTOX® 2 hours after Raltegravir in treatment period 4, followed by MINTOX® 2 hours before Raltegravir in treatment period 5. There was a minimum 2-day washout between treatment periods.
  Interventions: Drug: Raltegravir; Drug: TUMS® Ultra Strength; Drug: MINTOX® Maximum Strength

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400 mg oral tablet taken with 240 mL water every 12 hours
  Throughout the study, participants will continue to take raltegravir along with their other HIV medications. On the day of co-dosing and intensive pharmacokinetic (PK) sampling, raltegravir will be dosed in the morning in a fasted state in all periods.
  Other Names: RAL; ISENTRESS™; MK-0518
Drug: TUMS® Ultra Strength — 3 tablets TUMS® Ultra Strength (US) 1000 mg
  Throughout the study, participants will continue to take raltegravir every 12 hours along with their other HIV medications. There will be a minimum of 2 days washout between treatment periods. On the day of co-dosing and intensive PK sampling, raltegravir will be dosed in the morning in a fasted state in all periods.
  Other Names: TUMS; calcium carbonate antacid
Drug: MINTOX® Maximum Strength — 20 mL MINTOX® Maximum Strength (MS)
  Throughout the study, participants will continue to take raltegravir every 12 hours along with their other HIV medications. There will be a minimum of 2 days washout between treatment periods. On the day of co-dosing and intensive PK sampling, raltegravir will be dosed in the morning in a fasted state in all periods.
  Other Names: MINTOX; magnesium/aluminum hydroxide antacid

SUMMARY:
This study will evaluate: (1) the effect of co-administration of single doses of calcium carbonate antacid and magnesium/aluminum hydroxide antacid on the steady-state plasma pharmacokinetic profile of raltegravir in human immunodeficiency virus (HIV)-infected participants; and (2) the effect of staggered dosing of a single dose of a magnesium/aluminum hydroxide antacid 2 hours before and 2 hours after administration of raltegravir on the steady-state plasma pharmacokinetic profile of raltegravir in the same participants.

The study will determine whether (1) the C12hrs of steady-state raltegravir after co-administration of single doses of calcium carbonate antacid is decreased to a clinically meaningful degree compared with C12hrs after administration of raltegravir alone; and whether (2) the C12hrs of steady-state raltegravir after co-administration of a single dose of magnesium/aluminum hydroxide antacid is decreased to a clinically meaningful degree compared with the C12hrs after administration of raltegravir alone.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected participant on a stable raltegravir dose (400 mg every 12 hours) as part of a stable anti-retroviral regimen (ARV) for at least 1 month and will maintain current ARV therapy throughout the study
* Body Mass Index ≤32 kg/m^2
* Good general health
* Can be a current smoker and/or user of nicotine or nicotine-containing products, but use of nicotine-containing products will not be permitted during the stay at the clinical research site

Exclusion Criteria:

* History of gastric bypass surgery
* Pregnant or nursing
* Mentally or legally incapacitated, has significant emotional problems, or has a history of a clinically significant psychiatric disorder; participants who have had situational depression may be enrolled at the discretion of the investigator.
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases (excluding HIV); participants with a history of uncomplicated kidney stones or childhood asthma may be enrolled at the discretion of the investigator.
* Active neoplastic disease deemed unstable or progressing by the investigator
* Currently taking rifampin or unable to refrain from use of any proton pump inhibitor and any histamine-2 (H2)-blockers, over-the-counter antacids, calcium supplements, or multivitamins during the study
* Consumes excessive amounts of alcohol
* Consumes excessive amounts of coffee, tea, cola, or other caffeinated beverages
* Major surgery or blood donation within the past 4 weeks
* History of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Regular user of any illicit drugs or history of drug (including alcohol) abuse within the past 6 months; current methadone or suboxone use is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kiser JJ, Bumpass JB, Meditz AL, Anderson PL, Bushman L, Ray M, Predhomme JA, Rower J, Mawhinney S, Brundage R. Effect of antacids on the pharmacokinetics of raltegravir in human immunodeficiency virus-seronegative volunteers. Antimicrob Agents Chemother. 2010 Dec;54(12):4999-5003. doi: 10.1128/AAC.00636-10. Epub 2010 Oct 4. PMID 20921313

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | RAL, TUMS+RAL, MINTOX+RAL, MINTOX Before RAL, MINTOX After RAL | TUMS+RAL, MINTOX+RAL, RAL, MINTOX Before RAL, MINTOX After RAL | MINTOX+RAL, RAL, TUMS+RAL, MINTOX Before RAL, MINTOX After RAL | RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL | TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL | MINTOX+RAL, TUMS+RAL, RAL, MINTOX After RAL, MINTOX Before RAL
Started | 4 | 5 | 4 | 6 | 4 | 4
Completed | 4 | 4 | 4 | 5 | 4 | 4
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | RAL, TUMS+RAL, MINTOX+RAL, MINTOX Before RAL, MINTOX After RAL | TUMS+RAL, MINTOX+RAL, RAL, MINTOX Before RAL, MINTOX After RAL | MINTOX+RAL, RAL, TUMS+RAL, MINTOX Before RAL, MINTOX After RAL | RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL | TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL | MINTOX+RAL, TUMS+RAL, RAL, MINTOX After RAL, MINTOX Before RAL
Started | 4 | 4 | 4 | 5 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 3
Arm/Group | RAL, TUMS+RAL, MINTOX+RAL, MINTOX Before RAL, MINTOX After RAL | TUMS+RAL, MINTOX+RAL, RAL, MINTOX Before RAL, MINTOX After RAL | MINTOX+RAL, RAL, TUMS+RAL, MINTOX Before RAL, MINTOX After RAL | RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL | TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL | MINTOX+RAL, TUMS+RAL, RAL, MINTOX After RAL, MINTOX Before RAL
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 3 | 4 | 4 | 4 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | RAL, TUMS+RAL, MINTOX+RAL, MINTOX Before RAL, MINTOX After RAL | TUMS+RAL, MINTOX+RAL, RAL, MINTOX Before RAL, MINTOX After RAL | MINTOX+RAL, RAL, TUMS+RAL, MINTOX Before RAL, MINTOX After RAL | RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL | TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL | MINTOX+RAL, TUMS+RAL, RAL, MINTOX After RAL, MINTOX Before RAL
Started | 4 | 3 | 4 | 4 | 4 | 4
Completed | 4 | 3 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | RAL, TUMS+RAL, MINTOX+RAL, MINTOX Before RAL, MINTOX After RAL | TUMS+RAL, MINTOX+RAL, RAL, MINTOX Before RAL, MINTOX After RAL | MINTOX+RAL, RAL, TUMS+RAL, MINTOX Before RAL, MINTOX After RAL | RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL | TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL | MINTOX+RAL, TUMS+RAL, RAL, MINTOX After RAL, MINTOX Before RAL
Started | 4 | 3 | 4 | 4 | 4 | 4
Completed | 4 | 3 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL: Participants received MINTOX® + Raltegravir in treatment period 1, followed by Raltegravir in treatment period 2, followed by TUMS® + Raltegravir in treatment period 3, followed by MINTOX® 2 hours before Raltegravir in treatment period 4, followed by MINTOX® 2 hours after Raltegravir in treatment period 5. There was a minimum 2-day washout between treatment periods.
- TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL: Participants received Raltegravir in treatment period 1, followed by MINTOX® + Raltegravir in treatment period 2, followed by TUMS® + Raltegravir in treatment period 3, followed by MINTOX® 2 hours after Raltegravir in treatment period 4, followed by MINTOX® 2 hours before Raltegravir in treatment period 5. There was a minimum 2-day washout between treatment periods.
- Total: Total of all reporting groups
Arm/Group | RAL, TUMS+RAL, MINTOX+RAL, MINTOX Before RAL, MINTOX After RAL | TUMS+RAL, MINTOX+RAL, RAL, MINTOX Before RAL, MINTOX After RAL | MINTOX+RAL, RAL, TUMS+RAL, MINTOX Before RAL, MINTOX After RAL | RAL, MINTOX+RAL, TUMS+RAL, MINTOX After RAL, MINTOX Before RAL | TUMS+RAL, RAL, MINTOX+RAL, MINTOX After RAL, MINTOX Before RAL | MINTOX+RAL, TUMS+RAL, RAL, MINTOX After RAL, MINTOX Before RAL | Total
Number analyzed (Participants) | 4 | 5 | 4 | 6 | 4 | 4 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (10.4) | 46.6 (9.5) | 36.8 (15.4) | 40.3 (10.3) | 39.8 (11.8) | 40.8 (11.6) | 41.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 2 | 0 | 0 | 5
  Male | 2 | 4 | 4 | 4 | 4 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Steady State Plasma Concentration (C12hrs) of Raltegravir After Coadministration of Antacid (Primary Hypothesis)
Description: Participant blood samples were collected to measure the steady state plasma concentration of raltegravir 12 hours after administration alone or with a single dose of antacid. The primary hypothesis compared C12hrs of raltegravir when administered alone with C12hrs of raltegravir when coadministered with TUMS® or MINTOX®.
Time Frame: 12 hours postdose
Population: All participants were included for whom at least one pharmacokinetic (PK) parameter could be calculated for all treatment periods and who did not have any protocol deviation interfering with pharmacokinetics
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Groups:
- Raltegravir: Raltegravir 400 mg every 12 hours
- TUMS® + Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of TUMS® 1000 mg (3 tablets) was coadministered with raltegravir on the day of pharmacokinetic (PK) sampling
- MINTOX® + Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of MINTOX® 20 mL was coadministered with raltegravir on the day of PK sampling
Arm/Group | Raltegravir | TUMS® + Raltegravir | MINTOX® + Raltegravir
Number analyzed (Participants) | 26 | 24 | 25
nM | 132.30 (112) [101.14 to 173.05] | 89.75 (134) [68.08 to 118.32] | 49.38 (32.6) [37.62 to 64.81]
Statistical Analysis 1: Comparison: Raltegravir vs TUMS® + Raltegravir; Test type: Non-Inferiority or Equivalence — The hypothesis will be supported if the lower limit of the 90% confidence interval (CI) falls above 0.4 for the geometric least squares mean ratio for TUMS® + raltegravir versus raltegravir alone; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and treatment period and random effect for participant; Geometric Least Squares Mean Ratio = 0.678, 90% CI 2-sided [0.531 to 0.866] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean C12hrs for TUMS® + raltegravir / geometric least squares mean C12hrs for raltegravir alone
Statistical Analysis 2: Comparison: Raltegravir vs MINTOX® + Raltegravir; Test type: Non-Inferiority or Equivalence — The hypothesis will be supported if the lower limit of the 90% CI falls above 0.4 for the geometric least squares mean ratio for MINTOX® + raltegravir versus raltegravir alone; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and treatment period and random effect for participant; Geometric Least Squares Mean Ratio = 0.373, 90% CI 2-sided [0.293 to 0.475] — The parameter estimated, geometric least squares mean ratio, is the geometric least squares mean C12hrs for MINTOX® + raltegravir / geometric least squares mean C12hrs for raltegravir alone

2. Primary Outcome: Least Squares Mean Steady State Plasma Concentration (C12hrs) of Raltegravir After Staggered Administration of Antacid (Secondary Hypothesis)
Description: Participant blood samples were collected to measure the steady state plasma concentration of raltegravir 12 hours after administration alone or before or after a single dose of antacid. The secondary hypothesis compared C12hrs of raltegravir when administered alone with C12hrs of raltegravir when administered 2 hours before or after MINTOX®.
Time Frame: 12 hours postdose
Population: All participants were included for whom at least one PK parameter could be calculated for all treatment periods and who did not have any protocol deviation interfering with pharmacokinetics
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Groups:
- MINTOX® Before Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of MINTOX® 20 mL was administered 2 hours before raltegravir on the day of PK sampling
- MINTOX® After Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of MINTOX® 20 mL was administered 2 hours after raltegravir on the day of PK sampling
Arm/Group | Raltegravir | MINTOX® Before Raltegravir | MINTOX® After Raltegravir
Number analyzed (Participants) | 26 | 23 | 23
nM | 125.75 [94.33 to 167.62] | 54.92 [41.36 to 72.91] | 54.47 [40.95 to 72.46]
Statistical Analysis 1: Comparison: Raltegravir vs MINTOX® Before Raltegravir; Test type: Non-Inferiority or Equivalence — The hypothesis will be supported if the lower limit of the 90% confidence interval (CI) falls above 0.4 for the geometric least squares mean ratio for MINTOX® before raltegravir versus raltegravir alone; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and random effect for participant; Geometric Least Squares Mean Ratio = 0.437, 90% CI 2-sided [0.344 to 0.554] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean C12hrs for MINTOX® before raltegravir / geometric least squares mean C12hrs for raltegravir alone
Statistical Analysis 2: Comparison: Raltegravir vs MINTOX® After Raltegravir; Test type: Non-Inferiority or Equivalence — The hypothesis will be supported if the lower limit of the 90% confidence interval (CI) falls above 0.4 for the geometric least squares mean ratio for MINTOX® after raltegravir versus raltegravir alone; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and random effect for participant; Geometric Least Squares Mean Ratio = 0.433, 90% CI 2-sided [0.341 to 0.550] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean C12hrs for MINTOX® after raltegravir / geometric least squares mean C12hrs for raltegravir alone

3. Primary Outcome: Least Squares Mean Steady State Area Under the Plasma Concentration-time Curve (AUC0-12hrs) of Raltegravir After Coadministration of Antacid (Primary Hypothesis)
Description: Participant blood samples were collected to measure the steady state AUC of raltegravir up to 12 hours after administration alone or with a single dose of antacid. The primary hypothesis compared AUC0-12hrs of raltegravir when administered alone with AUC0-12hrs of raltegravir when coadministered with TUMS® or MINTOX®.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nM*hr
Groups:
- TUMS® + Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of TUMS® 1000 mg (3 tablets) was coadministered with raltegravir on the day of PK sampling
Arm/Group | Raltegravir | TUMS® + Raltegravir | MINTOX® + Raltegravir
Number analyzed (Participants) | 26 | 24 | 25
nM*hr | 16399.76 (12300) [12728.79 to 21129.44] | 7294.30 (6690) [5613.53 to 9478.31] | 8358.67 (5040) [6456.83 to 10820.68]
Statistical Analysis 1: Comparison: Raltegravir vs TUMS® + Raltegravir; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and treatment period and random effect for participant; Geometric Least Squares Mean Ratio = 0.445, 90% CI 2-sided [0.350 to 0.565] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean AUC0-12hrs for TUMS® + raltegravir / geometric least squares mean AUC0-12hrs for raltegravir alone
Statistical Analysis 2: Comparison: Raltegravir vs MINTOX® + Raltegravir; Test type: Non-Inferiority or Equivalence — The hypothesis will be supported if the lower limit of the 90% confidence interval (CI) falls above 0.4 for the geometric least squares mean ratio for MINTOX® + raltegravir versus raltegravir alone; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and treatment period and random effect for participant; Geometric Least Squares Mean Ratio = 0.510, 90% CI 2-sided [0.402 to 0.646] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean AUC0-12hrs for MINTOX® + raltegravir / geometric least squares mean AUC0-12hrs for raltegravir alone

4. Primary Outcome: Least Squares Mean Steady State Area Under the Plasma Concentration-Time (AUC0-12hrs) of Raltegravir After Staggered Administration of Antacid (Secondary Hypothesis)
Description: Participant blood samples were collected to measure the steady state AUC of raltegravir up to 12 hours after administration alone or before or after a single dose of antacid. The secondary hypothesis compared AUC0-12hrs of raltegravir when administered alone with AUC0-12hrs of raltegravir when administered 2 hours before or after MINTOX®.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nM*hr
Arm/Group | Raltegravir | MINTOX® Before Raltegravir | MINTOX® After Raltegravir
Number analyzed (Participants) | 26 | 23 | 23
nM*hr | 17577.15 [13353.74 to 23136.29] | 8521.95 [5572.42 to 13032.70] | 12226.11 [7988.11 to 18712.53]
Statistical Analysis 1: Comparison: Raltegravir vs MINTOX® Before Raltegravir; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and random effect for participant; Geometric Least Squares Mean Ratio = 0.485, 90% CI 2-sided [0.351 to 0.669] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean AUC0-12hrs for MINTOX® before raltegravir / geometric least squares mean AUC0-12hrs for raltegravir alone
Statistical Analysis 2: Comparison: Raltegravir vs MINTOX® After Raltegravir; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and random effect for participant; Geometric Least Squares Mean Ratio = 0.696, 90% CI 2-sided [0.504 to 0.960] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean AUC0-12hrs for MINTOX® after raltegravir / geometric least squares mean AUC0-12hrs for raltegravir alone

5. Primary Outcome: Least Squares Mean Maximum Plasma Concentration (Cmax) of Raltegravir After Coadministration of Antacid (Primary Hypothesis)
Description: Participant blood samples were collected to measure the steady state maximum plasma concentration of raltegravir when administered alone or with a single dose of antacid. The primary hypothesis compared Cmax of raltegravir when administered alone with Cmax of raltegravir when coadministered with TUMS® or MINTOX®.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Raltegravir | TUMS® + Raltegravir | MINTOX® + Raltegravir
Number analyzed (Participants) | 26 | 24 | 25
nM | 5427.15 (4530) [4132.93 to 7126.66] | 2584.78 (1700) [1949.15 to 3427.70] | 3013.88 (1940) [2282.54 to 3979.54]
Statistical Analysis 1: Comparison: Raltegravir vs TUMS® + Raltegravir; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and treatment period and random effect for participant; Geometric Least Squares Mean Ratio = 0.476, 90% CI 2-sided [0.362 to 0.627] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean Cmax for TUMS® + raltegravir / geometric least squares mean Cmax for raltegravir alone
Statistical Analysis 2: Comparison: Raltegravir vs MINTOX® + Raltegravir; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and treatment period and random effect for participant; Geometric Least Squares Mean Ratio = 0.555, 95% CI 2-sided [0.423 to 0.729] — The parameter estimated, geometric least squares mean ratio, is the geometric least squares mean Cmax for MINTOX® + raltegravir / geometric least squares mean Cmax for raltegravir alone

6. Primary Outcome: Least Squares Mean Maximum Plasma Concentration (Cmax) of Raltegravir After Staggered Administration of Antacid (Secondary Hypothesis)
Description: Participant blood samples were collected to measure the maximum steady state plasma concentration of raltegravir after administration alone or before or after a single dose of antiacid. The secondary hypothesis compared Cmax of raltegravir when administered alone with Cmax of raltegravir when administered 2 hours before or after MINTOX®.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | Raltegravir | MINTOX® Before Raltegravir | MINTOX® After Raltegravir
Number analyzed (Participants) | 26 | 23 | 23
nM | 5678.90 [4263.73 to 7563.78] | 2753.64 [1689.26 to 4488.68] | 4399.66 [2698.18 to 7174.09]
Statistical Analysis 1: Comparison: Raltegravir vs MINTOX® Before Raltegravir; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and random effect for participant; Geometric Least Squares Mean Ratio = 0.485, 90% CI 2-sided [0.332 to 0.709] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean Cmax for MINTOX® before raltegravir / geometric least squares mean Cmax for raltegravir alone
Statistical Analysis 2: Comparison: Raltegravir vs MINTOX® After Raltegravir; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Mixed Models Analysis; Analysis incorporated fixed effect for treatment and random effect for participant; Geometric Least Squares Mean Ratio = 0.775, 90% CI 2-sided [0.530 to 1.132] — The parameter estimated, geometric least squares mean ratio, is geometric least squares mean Cmax for MINTOX® after raltegravir / geometric least squares mean Cmax for raltegravir alone

7. Primary Outcome: Mean Time to Maximum Plasma Concentration (Tmax) of Raltegravir
Description: Participant blood samples were collected to measure the time to achieve the maximum steady state plasma concentration of raltegravir when administered alone or with a single dose of antacid
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Raltegravir | TUMS® + Raltegravir | MINTOX® + Raltegravir | MINTOX® Before Raltegravir | MINTOX® After Raltegravir
Number analyzed (Participants) | 26 | 24 | 25 | 23 | 23
hr | 2.06 (1.23) | 2.08 (1.64) | 1.48 (0.94) | 1.52 (1.17) | 1.78 (1.37)

8. Primary Outcome: Number of Participants With Any Clinical or Laboratory Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the
  structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an adverse experience.
Time Frame: Up to 7 days after the last dose of study drug
Population: All subjects who received any amount of the study drug were included in the safety population
Measure: Number; unit: participants
Groups:
- TUMS® + Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of TUMS® 1000 mg (3 tablets) was coadministered with raltegravir on the day of AE assessment
- MINTOX® + Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of MINTOX® 20 mL was coadministered with raltegravir on the day of AE assessment
- MINTOX® Before Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of MINTOX® 20 mL was administered 2 hours before raltegravir on the day of AE assessment
- MINTOX® After Raltegravir: Raltegravir 400 mg every 12 hours. A single dose of MINTOX® 20 mL was administered 2 hours after raltegravir on the day of AE assessment
Arm/Group | Raltegravir | TUMS® + Raltegravir | MINTOX® + Raltegravir | MINTOX® Before Raltegravir | MINTOX® After Raltegravir
Number analyzed (Participants) | 26 | 25 | 25 | 23 | 23
participants | 1 | 2 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 7 days after the last dose of study drug
Description: All subjects who received any amount of the study drug were included in the safety population.
Arm/Group | Raltegravir | TUMS® + Raltegravir | MINTOX® + Raltegravir | MINTOX® Before Raltegravir | MINTOX® After Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.